CLINICAL TRIAL: NCT02644798
Title: Nucleotide Polymorphism in ARDS Outcome: a Whole Exome Sequencing Association Study
Brief Title: Nucleotide Polymorphism in ARDS Outcome
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Principal Investigator, Southeast University, China
Other Study IDs: 2015ZDSYLL014.0
Record Dates: First submitted 2015-04-20; First posted 2016-01-01 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: ARDS
Keywords: ARDS; Nucleotide polymorphism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARDS patients: Adult ARDS (according to Berlin definition) patients were enrolled in the trial. The diagnostic criteria included (a) within one week of a known clinical insult or new or worsening respiratory symptoms; (b) chest imaging showing that bilateral opacities-not fully explained by effusions, lobar/lung collapse, or nodules; (c) respiratory failure not fully explained by cardiac failure or fluid overload; and (d) arterial partial pressure of oxygen / fraction of inspiration oxygen (PaO2/FiO2 ratio, P/F ratio) less than or equal to 300 mmHg.
  Interventions: Other: Baseline-recorded data recorded

INTERVENTIONS:
Other: Baseline-recorded data recorded — Baseline-recorded data recorded. Peripheral blood samples were drawn.

SUMMARY:
Acute respiratory distress syndrome (ARDS) is characterized by increased pulmonary vascular permeability and reduced aerated lung tissue. With an extremely high hospital mortality among 35 - 46%, current therapeutic strategies to increase ARDS survival are still limited. Advances in etiology and pathology of ARDS are urging. Numerous genetic variants were identified associated with ARDS outcome. By whole-exome sequencing association study, our goal was to explore the associations between genetic variants and ARDS outcome.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is characterized by increased pulmonary vascular permeability and reduced aerated lung tissue. With an extremely high hospital mortality among 35 - 46%, current therapeutic strategies to increase ARDS survival are still limited. Advances in etiology and pathology of ARDS are urging. Numerous genetic variants were identified associated with ARDS outcome. Then a few genetic risk factors have been discovered by large-scale genotyping approaches, from in vivo or in vitro models of lung injury, which highlight the importance of identifying genetic biomarkers of ARDS outcome to further improve stratification. The mutational landscape and variability at single nucleotide polymorphisms (SNP) with ARDS outcome in Chinese is unknown, not to mention their associations. By whole-exome sequencing association study, our goal was to explore the associations between genetic variants and ARDS outcome.

ELIGIBILITY:
Inclusion Criteria:

Adult ARDS (according to Berlin definition) patients were enrolled in the trial.

The diagnostic criteria included

1. within one week of a known clinical insult or new or worsening respiratory symptoms;
2. chest imaging showing that bilateral opacities-not fully explained by effusions, lobar/lung collapse, or nodules;
3. respiratory failure not fully explained by cardiac failure or fluid overload;
4. arterial partial pressure of oxygen / fraction of inspiration oxygen (PaO2/FiO2 ratio, P/F ratio) less than or equal to 300 mmHg.

Exclusion criteria:

Patients refused to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS adult patients
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Number of survived participants | through study completion, an average of 28 day
  Survivors and non-survivors in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, M.D., Principal Investigator — Southeast University
Locations (1):
- Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Famous KR, Delucchi K, Ware LB, Kangelaris KN, Liu KD, Thompson BT, Calfee CS; ARDS Network. Acute Respiratory Distress Syndrome Subphenotypes Respond Differently to Randomized Fluid Management Strategy. Am J Respir Crit Care Med. 2017 Feb 1;195(3):331-338. doi: 10.1164/rccm.201603-0645OC. PMID 27513822
- [Result] Calfee CS, Janz DR, Bernard GR, May AK, Kangelaris KN, Matthay MA, Ware LB. Distinct molecular phenotypes of direct vs indirect ARDS in single-center and multicenter studies. Chest. 2015 Jun;147(6):1539-1548. doi: 10.1378/chest.14-2454. PMID 26033126
- [Result] Shankar-Hari M, McAuley DF. Acute Respiratory Distress Syndrome Phenotypes and Identifying Treatable Traits. The Dawn of Personalized Medicine for ARDS. Am J Respir Crit Care Med. 2017 Feb 1;195(3):280-281. doi: 10.1164/rccm.201608-1729ED. No abstract available. PMID 28145757
- [Result] Calfee CS, Delucchi K, Parsons PE, Thompson BT, Ware LB, Matthay MA; NHLBI ARDS Network. Subphenotypes in acute respiratory distress syndrome: latent class analysis of data from two randomised controlled trials. Lancet Respir Med. 2014 Aug;2(8):611-20. doi: 10.1016/S2213-2600(14)70097-9. Epub 2014 May 19. PMID 24853585
- [Derived] Xu JY, Liu AR, Wu ZS, Xie JF, Qu XX, Li CH, Meng SS, Liu SQ, Yang CS, Liu L, Huang YZ, Guo FM, Yang Y, Qiu HB. Nucleotide polymorphism in ARDS outcome: a whole exome sequencing association study. Ann Transl Med. 2021 May;9(9):780. doi: 10.21037/atm-20-5728. PMID 34268393